CLINICAL TRIAL: NCT03145350
Title: The Effect of a High Fat Compared to a High Sugar Diet on Liver Fat Accumulation and Metabolism
Brief Title: The Effect of a High-fat vs. High-sugar Diet on Liver Fat Accumulation and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Oxlip-2017-HFD/HSD
Record Dates: First submitted 2017-01-09; First posted 2017-05-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2018-05

CONDITIONS: Fat; Liver; NAFLD
Keywords: NAFLD; Fat intake; Sugar intake
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Randomised crossover with washout period.
Who Masked: Investigator
Masking Description: PI,and research assistants undertaking measurements will be blinded to the dietary intervention the participant is undertaking.
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-fat, low-carbohydrate diet (Active Comparator): Dietary intervention: Participants will consume a diet that is rich in saturated fat (20% total energy) and low in free sugars for 4 weeks. This diet will include commonly eaten foods such as butter, cheese, and fatty meat products. Total fat intake in this intervention will be 40-45% total energy.
  Interventions: Other: High-fat, low-carbohydrate
- Low-fat, high-carbohydrate diet (Active Comparator): Dietary intervention: Participants will consume a diet that is low in saturated fat (~5% total energy) and rich in free sugars (20% total energy).The diet will include commonly eaten food and drink such as sugar sweetened beverages, confectionery (e.g. fruit gums) and table sugar.
  Interventions: Other: Low-fat, high-carbohydrate

INTERVENTIONS:
Other: High-fat, low-carbohydrate — Dietary intervention: 4 week
  Arms: High-fat, low-carbohydrate diet
Other: Low-fat, high-carbohydrate — Dietary intervention: 4 week
  Arms: Low-fat, high-carbohydrate diet

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most prevalent liver disease in the world. It is currently unclear why fat starts to accumulate in the liver, although both the amount and type of food consumed have been implicated. The majority of studies that have investigated the effects of dietary fat or sugar on liver fat have fed volunteers excess calories, which are known to increase liver fat. The effect of specific dietary components, when consumed as part of a diet not containing excess calories, on liver fat accumulation remains unclear.

DETAILED DESCRIPTION:
This research aims to investigate the role excessive consumption of specific macronutrients may play in the development of NAFLD. This will be achieved by subjecting participants to two specific dietary interventions (high-fat, low-carbohydrate and low-fat, high-carbohydrate) in a randomized, crossover research design. Liver fat content, and whole-body and hepatic fasting and postprandial lipid metabolism will be assessed before and after the specific dietary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* BMI >25 <35kg/m2
* No medical condition or relevant drug therapy known to affect liver, lipid or glucose metabolism

Exclusion Criteria:

* Age <30 or >65 years
* Body mass index <25 or >35kg/m2
* A blood haemoglobin <120mg/dL
* Any metabolic condition or relevant drug therapy
* People who do not tolerate fructose
* Smoking
* History of alcoholism or a greater than recommended alcohol intake
* Pregnant or nursing mothers
* Women prescribed any contraceptive agent or device including oral contraceptives, hormone replacement therapy (HRT) or who have used these within the last 12 months
* History of severe claustrophobia
* Presence of metallic implants, pacemaker
* Haemorrhagic disorders
* Anticoagulant treatment

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content | Before, and within 7 days after completion of each dietary intervention
  Investigators will measure the change in liver fat content after each of the 4 week intervention diets by magnetic resonance imaging/spectroscopy (MRI/S).

SECONDARY OUTCOMES:
Change in hepatic fatty acid partitioning | Within 7 days after completion of each dietary intervention
  Investigators will utilise stable isotope tracer methodology to measure the contribution of newly synthesised fatty acids and dietary fatty acids to triglyceride production and oxidation pathways in the liver after each of the 4 week intervention diets.
Change in plasma metabolite concentrations | Before, and within 7 days after completion of each dietary intervention.
  Circulating concentrations of glucose, insulin, non-esterified fatty acids, and triglycerides will be measured biochemically using a clinical analyser after each of the 4 week intervention diets.
Change in whole-body fatty acid oxidation | Within 7 days after completion of each dietary intervention
  Investigators will utilise stable isotope tracer methodology to measure whole-body dietary fatty acid oxidation after each of the 4 week intervention diets.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Hodson, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the study, all individual data obtained from participants may potentially be shared with other researchers, both here in the United Kingdom and abroad, in appropriate circumstances. If data is to be shared with other researchers, it will be done so under fully anonymised conditions.

REFERENCES:
- [Derived] Parry SA, Rosqvist F, Mozes FE, Cornfield T, Hutchinson M, Piche ME, Hulsmeier AJ, Hornemann T, Dyson P, Hodson L. Intrahepatic Fat and Postprandial Glycemia Increase After Consumption of a Diet Enriched in Saturated Fat Compared With Free Sugars. Diabetes Care. 2020 May;43(5):1134-1141. doi: 10.2337/dc19-2331. Epub 2020 Mar 12. PMID 32165444